CLINICAL TRIAL: NCT00414167
Title: Placebo-Controlled Trial of Bupropion for the Treatment of Binge Eating Disorder
Brief Title: Craving, Binge Eating and Obesity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0511000832; K23DK071646 (NIH)
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Binge Eating Disorder; Obesity
Keywords: Binge eating; Obesity; Medication; Craving; Emotional eating
MeSH Terms: conditions — Binge-Eating Disorder; Obesity; Bulimia; Emotional Eating | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Bupropion
  Interventions: Drug: bupropion
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: bupropion — 300 mg per day for 8 weeks
  Other Names: wellbutrin; zyban
  Arms: 1
Other: Placebo — Placebo
  Arms: 2

SUMMARY:
This research study is designed to look at the effectiveness of bupropion for reducing binge eating in overweight persons with binge eating problems. Participants in the study will receive either bupropion or placebo ("sugar" pill, inactive medication) as an outpatient for eight weeks. In addition, participants will be given the option to receive 8 weeks of free behavioral weight loss treatment. This treatment, known to be effective for reducing binge eating and helping people lose weight, will be administered following the medication phase and at no cost.

It is expected that compared to placebo, bupropion will produce greater reductions in binge eating.

DETAILED DESCRIPTION:
The proposed study is an 8-week randomized placebo-controlled trial to test the efficacy of bupropion in treating overweight women with binge eating disorder (BED). Bupropion is an antidepressant that has demonstrated efficacy in smoking cessation and some efficacy in obesity treatment. Since cravings and depressed mood are hypothesized to contribute to binge eating episodes, bupropion is a promising psychopharmacological agent in treating binge eating and reducing weight. It is hypothesized that compared to placebo, bupropion will produce significantly greater reductions in the frequency of binge eating. Secondary goals are to explore interrelationships between treatment and changes in cravings, frequency of binge episodes, emotional eating, and weight loss. Following the medication phase of the trial, all patients will be offered 8 weeks of behavioral weight loss treatment administered by doctoral-level psychologists specializing in eating disorders and weight management.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-50
* Able to travel to clinical site (New Haven, CT) for bi-weekly visits.

Exclusion Criteria:

* Predisposition to seizures
* History of anorexia or bulimia nervosa
* Current Type I or Type II diabetes mellitus

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marney A. White, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] White MA, Grilo CM. Bupropion for overweight women with binge-eating disorder: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2013 Apr;74(4):400-6. doi: 10.4088/JCP.12m08071. PMID 23656848

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-one overweight and obese women with BED were recruited from the community via advertisements. Participants were enrolled from November 2006 to December 2010. Assessments and clinic appointments were held in a medical school research clinic.
Groups:
- Bupropion (300 mg/d): Bupropion
  bupropion : 300 mg per day for 8 weeks
- Placebo: Placebo
  Placebo : Placebo
Period: Overall Study
Arm/Group | Bupropion (300 mg/d) | Placebo
Started | 31 | 30
Completed | 27 | 27
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Bupropion: Bupropion
  bupropion : 300 mg per day for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Bupropion | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.1) | 43.1 (13.0) | 44.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Binge Eating Episodes
Time Frame: One week (at post treatment)
Population: Baseline forward imputation for missing data.
Measure: Mean (Standard Deviation); unit: episodes/week
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 31 | 30
episodes/week | 0.8 (1.2) | 1.0 (1.5)

2. Secondary Outcome: Percent BMI Loss
Description: Percent loss in Body Mass Index
Time Frame: 8 weeks (baseline and 8 weeks)
Population: Baseline values imputed forward for missing data.
Measure: Mean (Standard Deviation); unit: Percent loss
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 31 | 20
Percent loss | 1.8 (2.6) | 0.6 (2.1)

ADVERSE EVENTS:
Arm/Group | Bupropion | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No